CLINICAL TRIAL: NCT00263835
Title: A Self-care Intervention for Latino Adults With Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK59527 (completed); 5R01DK059527-04 (NIH)
Record Dates: First submitted 2005-12-07; First posted 2005-12-09 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

INTERVENTIONS:
Behavioral: Empowerment

SUMMARY:
The purpose of this study is to modify and evaluate a culturally appropriate intervention that is designed to improve diabetes self-care practices by enhancing the self-efficacy, empowerment and diabetes knowledge among Latino adults over the age of 55 years.

DETAILED DESCRIPTION:
It is recognized that Latinos with diabetes experience substantially worse process and outcomes of care. To address this problem, the goal of the proposed study is to modify and evaluate a culturally appropriate intervention designed to improve diabetes self-care practices by enhancing the self-efficacy, empowerment, and diabetes-specific knowledge among Latino adults over the age of 55 years. Specific aims of the project are: 1) to modify an existing empowerment intervention to improve self-care skills among Latinos with diabetes; 2) to test the effect of a patient-centered culturally-tailored intervention that focuses on increasing self-efficacy, knowledge about diabetes care, and self-care skills among Latinos with diabetes on: a) biophysiological endpoints such as glycemic control; b) self-efficacy, diabetes-specific knowledge, and self-care behaviors; c) psychosocial endpoints such as quality of life; and d) total costs and cost-effectiveness of care; and 3) to test the effect of the intervention on compliance with indicators of good process of diabetes care. To evaluate the effectiveness of the intervention, the research team will conduct a controlled clinical trial that will randomize 300 Latino adults over the age of 55 years with diabetes who are cared for in 4 public clinics affiliated with the Martin Luther King/Drew University Medical Center. Randomization will occur at the patient level. The primary endpoints for the trial will be: 1) differences in glycemic control as reflected by mean difference in hemoglobin A1c over time for the intervention versus usual care control group; and 2) difference in diabetes-specific quality of life over time. The trial will also measure a number of important secondary endpoints both before and after exposure to the intervention: self-efficacy, knowledge about diabetes, self-care behaviors, diabetes-specific symptoms, quality of life, low density lipoprotein levels, blood pressure, weight, quality of care, and costs. Variables that are likely to modify the effectiveness of the intervention will also be examined, including acculturation, language, insurance status, and social support. These data will provide the needed information to evaluate both the effectiveness and the cost effectiveness of the patient-centered intervention among Latino adults with diabetes. In summary, by modifying and testing an empowerment intervention that focuses on the patient, we hope to arm Latino adults with diabetes with the needed self-efficacy, knowledge, and self-care skills to have the best possible glycemic control and process of health care regardless of the resources available in their care setting.

ELIGIBILITY:
Inclusion Criteria:

Self-Identify as having diabetes, be 55 years of age or older, Latino/a and have a hemoglobing A1c of 8% or greater.

Exclusion Criteria:

Non diabetic, under 55, non Latino/a, a hemoglobin A1c of less than 8%.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-10; Study Completion 2006-05

PRIMARY OUTCOMES:
Change in hemoglobin A1c.

SECONDARY OUTCOMES:
Change in blood pressure, cholesterol, and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Carol M Mangione, M.D., MSPH, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Derived] Sugiyama T, Steers WN, Wenger NS, Duru OK, Mangione CM. Effect of a community-based diabetes self-management empowerment program on mental health-related quality of life: a causal mediation analysis from a randomized controlled trial. BMC Health Serv Res. 2015 Mar 22;15:115. doi: 10.1186/s12913-015-0779-2. PMID 25880234